CLINICAL TRIAL: NCT05780463
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With COVID-19 (Trial H5: MP0420)
Brief Title: MP0420 for Inpatients With COVID-19 (An ACTIV-3/TICO Treatment Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Molecular Partners AG (Industry); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 014/ACTIV-3/H5
Record Dates: First submitted 2023-03-20; First posted 2023-03-22 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3; TICO
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — ensovibep; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MP0420 plus SOC (Experimental): * MP0420 600 mg solution (4 vials of 15 mg/mL); administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Drug: MP0420; Biological: Remdesivir
- Placebo plus SOC (Placebo Comparator): * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Drug: Placebo; Biological: Remdesivir

INTERVENTIONS:
Drug: MP0420 — MP0420 is a multi-valent DARPin® molecule (designed ankyrin repeat protein), consisting of 5 DARPin® domains.
  Other Names: ensovibep
  Arms: MP0420 plus SOC
Drug: Placebo — Commercially available 0.9% sodium chloride solution
  Arms: Placebo plus SOC
Biological: Remdesivir — Antiviral agent
  Other Names: Veklury

SUMMARY:
This study looks at the safety and effectiveness of MP0420 in treating COVID-19 in people who have been hospitalized with the infection. Participants in the study will be treated with either MP0420 plus current standard of care (SOC), or with placebo plus current SOC. This is ACTIV-3/TICO Treatment Trial H5.

DETAILED DESCRIPTION:
This is a treatment trial of the ACTIV-3/TICO master protocol (NCT04501978) to evaluate the safety and efficacy of MP0420 in hospitalized patients infected with COVID-19.

This is a randomized, blinded, controlled sub-study of MP0420 plus current SOC against placebo plus current SOC. The placebo arm may be shared across other sub-studies of the ACTIV-3/TICO master protocol. When more than one drug is being tested at the same time, participants will be randomly allocated to treatments or placebo.

Randomization will be stratified by study site pharmacy and disease severity. There are 2 disease severity strata: participants without organ failure (severity stratum 1) and participants with organ failure (severity stratum 2).

An independent Data and Safety Monitoring Board (DSMB) will regularly review interim analyses and summarize safety and efficacy outcomes. The pace of enrollment with be initially restricted, and there will be an early review of safety data by the DSMB. At the outset of the trial, only participants in disease severity stratum 1 will be enrolled. This will continue until approximately 300 participants are enrolled and followed for 5 days. The exact number will vary according to the speed of enrollment and the timing of DSMB meetings. Prior to expanding enrollment to also include patients in disease severity stratum 2, safety will be evaluated and a pre-specified futility assessment by the DSMB will be carried out using 2 ordinal outcomes assessed at Day 5.

If MP0420 passes the futility assessment, enrollment of participants will be expanded, seamlessly and without any data unblinding, to include participants in disease severity stratum 2 as well as those in disease severity stratum 1. Future interim analyses will be based on the primary endpoint of sustained recovery and will use pre-specified guidelines to determine early evidence of benefit, harm, or futility for the investigational agent. Participants will be followed for 18 months following randomization.

This trial will be conducted in several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

ELIGIBILITY:
Inclusion Criteria: Refer to the master protocol (NCT04501978)

Exclusion Criteria: Refer to the master protocol (NCT04501978)

Additional Exclusion Criteria:

1. Pregnant women
2. Nursing mothers
3. Women of child-bearing potential who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with men or practice appropriate contraception through 11 weeks after receiving MP0420/placebo
4. Men who are unwilling to acknowledge the strong advice to abstain from sexual intercourse with women of child-bearing potential or to use barrier contraception through 11 weeks after receiving MP0420/placebo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Prof., Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen; James Neaton, Prof., Study Chair — INSIGHT Statistical and Data Management Center, University of Minnesota
Locations (105):
- United States (73):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - Southern Arizona VA Healthcare System (Site 074-009), 3601 S. 6th Ave., Tucson, Arizona
  - Velocity Chula Vista (Site 080-034), 752 Medical Center Ct., Ste. 304, Chula Vista, California
  - Community Regional Medical Center (Site 203-005), 2823 Fresno Street, Fresno, California
  - Velocity San Diego (Site 080-035), 5565 Grossmont Center Drive, Building 2, Suite 1, La Mesa, California
  - VA Long Beach Healthcare System (Site 074-026), 5901 East 7th Street (09/151-M2), Long Beach, California
  - Cedars-Sinai Medical Center (Site 208-002), 8700 Beverly Blvd., Los Angeles, California
  - Ronald Reagan UCLA Medical Center (Site 203-002), 757 Westwood Plaza, Los Angeles, California
  - Sacramento VA Medical Center (Site 074-023), 10535 Hospital Way, Mather, California
  - Hoag Memorial Hospital Presbyterian (Site 080-026), One Hoag Drive, Newport Beach, California
  - UC Davis Health (Site 203-004), 2315 Stockton Blvd., Sacramento, California
  - VA San Diego Healthcare System (Site 074-016), 3350 La Jolla Village Drive, San Diego, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - San Francisco VAMC (Site 074-002), 4150 Clement St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffitt-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Site 066-002), 1124 W. Carson Street, CDCRC Building, Torrance, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Public Health (Site 017-004), 660 Bannock St., MC2600 (Infectious Disease Clinic), Denver, Colorado
  - West Haven VA Medical Center (Site 025-007), 950 Campbell Avenue, West Haven, Connecticut
  - MedStar Health Research Institute (Site 009-021), MedStar Washington Hospital Center, 110 Irving St., NW., Washington D.C., District of Columbia
  - Washington DC VA Medical Center (Site 009-004), 50 Irving Street NW, Washington D.C., District of Columbia
  - Bay Pines VAMC (Site 074-004), 10000 Bay Pines Blvd., Bldg. 100, Room 5B-104, Bay Pines, Florida
  - Miami VAMC (Site 074-003), 1201 NW 16 Street, Miami, Florida
  - Hillsborough County Health Department, University of South Florida (Site 032-001), Tampa, Florida
  - Emory University (Site 301-008), The Emory Clinic, Bldg. A, Suite 2236, 1365 Clifton Rd., NE, Atlanta, Georgia
  - Lutheran Medical Group (Site 301-010), 7916 W. Jefferson Boulevard, Fort Wayne, Indiana
  - Cotton O'Neil Clinical Research Center (Site 080-030), Stormont Vail Health, 1500 SW 10th Avenue, Topeka, Kansas
  - Ochsner Clinic Foundation (Site 301-015), 1514 Jefferson Highway, New Orleans, Louisiana
  - University of Maryland Medical Center (Site 301-019), 22 South Greene Street, Baltimore, Maryland
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Site 202-001), 330 Brookline Ave., Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), 759 Chestnut Street, Springfield, Massachusetts
  - University of Michigan (Site 205-001), 1500 East Medical Center Drive, Ann Arbor, Michigan
  - Henry Ford Health System, Henry Ford Hospital (Site 014-001), 2799 W. Grand Blvd., Detroit, Michigan
  - Minneapolis Heart Institute Foundation (Site 301-026), Abbott Northwestern Hospital, 920 E 28th St. #100, Minneapolis, Minnesota
  - Hennepin Healthcare (Site 027-001), 701 Park Avenue, Minneapolis, Minnesota
  - Minneapolis VA Health Care System (Site 105-001), 1 Veterans Drive, Bldg 70, Minneapolis, Minnesota
  - M Health Fairview University of Minnesota Medical Center (Site 112-001), 500 Harvard St. SE., Minneapolis, Minnesota
  - University of Mississippi Medical Center (Site 202-005), 2500 North State Street, Jackson, Mississippi
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital (Site 301-024), One Medical Center Drive, Lebanon, New Hampshire
  - Cooper University Hospital (Site 019-001), One Cooper Plaza, Camden, New Jersey
  - SUNY Downstate Medical Center (Site 033-001), 450 Clarkson Ave., Brooklyn, New York
  - Maimonides Medical Center (Site 033-002), 4802 10th Avenue, Brooklyn, New York
  - Lincoln Medical Center (New York Health and Hospitals/Lincoln) (Site 003-016), 234 E. 149th Street, The Bronx, New York
  - Montefiore Medical Center Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest University Health Sciences (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center (Site 207-003), 234 Goodman Ave., Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center (Site 108-001), 11100 Euclid Avenue, Cleveland, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - Portland VA Healthcare System (Site 074-024), 3710 SW. US Veterans Hospital Road, Portland, Oregon
  - Rhode Island Hospital (Site 080-036), 593 Eddy Street, Providence, Rhode Island
  - The Miriam Hospital (Site 080-039), 164 Summit Ave., Providence, Rhode Island
  - Ralph H. Johnson VA Medical Center (Site 074-015), 109 Bee Street, Charleston, South Carolina
  - MUSC Research Nexus Clinic (Site 210-002), 96 Jonathan Lucas St., CSB 214, Charleston, South Carolina
  - MUSC Health Florence Medical Center (Site 210-006), 805 Pamplico Highway, Florence, South Carolina
  - VA TVHS Nashville Campus (Site 074-022), 1310 24th Avenue South, Nashville, Tennessee
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - Hendrick Medical Center (Site 080-014), 1900 Pine Street, Abilene, Texas
  - CHRISTUS Spohn Shoreline Hospital (Site 080-001), 600 Elizabeth Street, Corpus Christi, Texas
  - Parkland Health and Hospital Systems (Site 084-002), 5200 Harry Hines Blvd, Dallas, Texas
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center (MEDV AMC) (Site 074-006), 2002 Holcombe Blvd., Houston, Texas
  - Texas Heart Institute (Site 301-017), 6770 Bertner, MC4-266, Houston, Texas
  - CHRISTUS Good Shepherd Medical Center (Site 080-031), 700 E. Marshall Ave., Longview, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Virginia Health Systems (Site 301-021), 1215 Lee Street, Charlottesville, Virginia
  - Carilion Roanoke Memorial Hospital (Site 080-018), 1906 Belleview Avenue, Roanoke, Virginia
  - Salem VA Medical Center (Site 074-014), 1970 Roanoke Blvd., Salem, Virginia
  - Swedish Hospital First Hill (Site 208-005), 747 Broadway, Seattle, Washington
  - West Virginia University (Site 301-023), One Medical Center Drive, Morgantown, West Virginia
- Denmark (10):
  - Aalborg Hospital (Site 625-005), Hobrovej 18, Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Department of Infectious Diseases, Palle Juul-Hensens Boulevard 99, Aarhus N
  - Bispebjerg Hospital (Site 625-013), Bispebjerg Bakke 23, Copenhagen
  - Righospitalet (Site 625-006), Blegdamsvej 9,, Copenhagen Ø
  - Herlev/Gentofte Hospital (Site 625-012), Medicinsk Afdeling, Herlev Ringvej 75, Herlev
  - Nordsjællands Hospital (Site 625-009), Dyrehavevej 29, Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases (Site 625-001), Kettegård allé 30, Hvidovre
  - Kolding Sygehus (Site 625-011), Medicinsk Afdeling, Sygehusvej 24, Kolding
  - Odense University Hospital (Site 625-004), Infektionsmedicinsk Forskningsenhed, J.B. Winsløwsgade 4, Odense
  - Zealand University Hospital, Roskilde (Site 625-010), Sygehusvej 10, Roskilde
- Greece (5):
  - Democritus University of Thrace (Site 635-021), University General Hospital of Alexandroupolis, Dragana, Alexandroupoli, Evros
  - Evangelismos COVID-19 Unit, (Site 635-020), 1st Dept. of Pulmonary and Critical Care Medicine, Evangelismos General Hospital, Dept., Ipsilantou 45-47, Athens
  - 1st Respiratory Medicine Dept., Athens University Medical School (Site 635-015), Athens Hospital for Diseases of the Chest "Sotiria Hospital", 152 Mesogeion Ave., Athens
  - 3rd Dept. of Medicine, Medical School, NKUA (Site 635-022), Sotiria General Hospital, 152 Mesogeion Ave., Athens
  - Attikon University General Hospital (Site 635-009), 4th Dept. of Internal Medicine, Medical School, National and Kapodistrian University of Athens, 1 Rimini St., Haidari, Athens
- Institute of Human Virology Nigeria (IHVN) (Site 612-601), Plot 252, Herbert Macaulay Way, Central Business District, Abuja, Nigeria
- Wojewódzki Szpital Zakazny (Site 625-302), Wolska 37, Warsaw, Poland
- Tan Tock Seng Hospital (Site 612-201), National Centre for Infectious Diseases (NCID), 11 Jalan Tan Tock Seng, Singapore, Singapore
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol (Site 626-003), Infectious Disease Unit, Second Floor, Building Maternal, Road Canyet s/n, Badalona, Barcelona
  - Hospital Universitari Arnau de Vilanova (Site 626-035), Av. Alcalde Rovira Roure 80, Lleida, Leida
  - Hospital Del Mar (Site 626-025), Paseo Maritimo 25-29, Barcelona
  - Hospital Clínic de Barcelona (Site 626-004), Carrer de Villaroel 170, Barcelona
- University Hospital Zurich (Site 621-201), Department of Infectious Diseases and Hospital Epidemiology, Raemistrasse 100, Zurich, Canton of Zurich, Switzerland
- Uganda (6):
  - MRC/UVRI and LSHTM Uganda Research Unit (Site 634-601), Entebbe Regional Referral Hospital, Entebbe
  - Gulu Regional Referral Hospital (Site 634-603), Laroo Division, PO Box 160, Gulu
  - Makerere University Lung Institute (Site 634-604), New Mulago Hospital Complex, Mulago Hill, Kampala
  - St. Francis Hospital, Nsambya (Site 634-607), Nsambya Road Nsambya Hill, P.O. Box 7146, Kampala
  - Lira Regional Referral Hospital (Site 634-605), Lira
  - Masaka Regional Referral Hospital (Site 634-606), MRC/UVRI and LSHTM Uganda Research Unit, Plot 6 Circle Road, PO Box 556, Masaka
- United Kingdom (3):
  - Royal Victoria Infirmary (Site 634-007), Queen Victoria Road, Newcastle upon Tyne, Northumbria
  - Royal Free Hospital (Site 634-006), Pond Street, Hampstead, London
  - Guy's and St. Thomas' NHS Foundation Trust (Site 634-011), London

REFERENCES:
- [Result] ACTIV-3/TICO Study Group; Barkauskas C, Mylonakis E, Poulakou G, Young BE, Vock DM, Siegel L, Engen N, Grandits G, Mosaly NR, Vekstein AM, Rogers R, Shehadeh F, Kaczynski M, Mylona EK, Syrigos KN, Rapti V, Lye DC, Hui DS, Leither L, Knowlton KU, Jain MK, Marines-Price R, Osuji A, Overcash JS, Kalomenidis I, Barmparessou Z, Waters M, Zepeda K, Chen P, Torbati S, Kiweewa F, Sebudde N, Almasri E, Hughes A, Bhagani SR, Rodger A, Sandkovsky U, Gottlieb RL, Nnakelu E, Trautner B, Menon V, Lutaakome J, Matthay M, Robinson P, Protopapas K, Koulouris N, Kimuli I, Baduashvili A, Braun DL, Gunthard HF, Ramachandruni S, Kidega R, Kim K, Hatlen TJ, Phillips AN, Murray DD, Jensen TO, Padilla ML, Accardi EX, Shaw-Saliba K, Dewar RL, Teitelbaum M, Natarajan V, Laverdure S, Highbarger HC, Rehman MT, Vogel S, Vallee D, Crew P, Atri N, Schechner AJ, Pett S, Hudson F, Badrock J, Touloumi G, Brown SM, Self WH, North CM, Ginde AA, Chang CC, Kelleher A, Nagy-Agren S, Vasudeva S, Looney D, Nguyen HH, Sanchez A, Weintrob AC, Grund B, Sharma S, Reilly CS, Paredes R, Bednarska A, Gerry NP, Babiker AG, Davey VJ, Gelijns AC, Higgs ES, Kan V, Matthews G, Thompson BT, Legenne P, Chandra R, Lane HC, Neaton JD, Lundgren JD. Efficacy and Safety of Ensovibep for Adults Hospitalized With COVID-19 : A Randomized Controlled Trial. Ann Intern Med. 2022 Sep;175(9):1266-1274. doi: 10.7326/M22-1503. Epub 2022 Aug 9. PMID 35939810

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 62 sites in 10 countries (Denmark, Greece, Nigeria, Poland, Singapore, Spain, Switzerland, Uganda, UK, USA). The first subject was enrolled on 11 Jun 2021 and the last subject was enrolled on 15 Nov 2021.
Groups:
- MP0420 Plus SOC: * MP0420 600 mg solution (4 vials of 15 mg/mL); administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  MP0420: MP0420 is a multi-valent DARPin® molecule (designed ankyrin repeat protein), consisting of 5 DARPin® domains.
  Remdesivir: Antiviral agent
- Placebo Plus SOC: * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Placebo: Commercially available 0.9% sodium chloride solution
  Remdesivir: Antiviral agent
Period: Overall Study
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Started | 247 | 238
Completed | 247 | 238
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC | Total
Number analyzed (Participants) | 247 | 238 | 485
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (14.9) | 56.6 (16.6) | 56.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 110 | 210
  Male | 147 | 128 | 275
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 38 | 79
  Not Hispanic or Latino | 206 | 200 | 406
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 14 | 15 | 29
  Black or African American | 61 | 58 | 119
  American Indian or Alaska Native | 1 | 0 | 1
  White | 138 | 128 | 266
  Native Hawaiian or Pacific Islander | 1 | 1 | 2
  More than one race | 1 | 4 | 5
  Other | 6 | 8 | 14
  Only ethnicity reported | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Recovery
Description: Sustained recovery defined as being discharged from the index hospitalization, followed by being alive and home for 14 consecutive days prior to Day 90.
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 247 | 238
Participants | 203 | 190

2. Primary Outcome: Number of Participants With an Ordinal Outcome on Day 5
Description: Ordinal outcome with 7 mutually exclusive categories
Time Frame: Status on Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 242 | 233
Participants
  7 = Death | 1 | 3
  6 = Invasive ventilation, ECMO, mechanical circulatory support, new renal replacement therapy | 16 | 10
  5 = Non-invasive ventilation or high flow oxygen | 46 | 45
  4 = Supplement oxygen (≥4 L/min or ≥4 L/min above baseline, but not high flow oxygen) | 40 | 30
  3 = Supplement oxygen (<4 L/min or <4 L/min above baseline, but not high flow oxygen) | 36 | 45
  2 = Limiting symptoms due to COVID-19, but no need of new or increased oxygen from baseline | 58 | 49
  1 = No limiting symptoms due to COVID-19 | 45 | 51

3. Secondary Outcome: Number of Participants Who Died From All Causes
Description: All-cause mortality
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 247 | 238
Participants | 30 | 35

4. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 5
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 5
Time Frame: Through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 247 | 238
Participants | 61 | 70

5. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 28
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 247 | 238
Participants | 85 | 97

6. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 90
Description: Death, SAE, clinical organ failure, serious infections through Day 90
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 247 | 238
Participants | 78 | 70

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Only Grade 3 or 4 AEs were collected.
Arm/Group | MP0420 Plus SOC | Placebo Plus SOC
All-Cause Mortality (participants affected / at risk) | 30/247 | 35/238
Serious Adverse Events (participants affected / at risk) | 14/247 | 18/238
Other Adverse Events (participants affected / at risk) | 65/247 | 79/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP0420 Plus SOC (N=247) | Placebo Plus SOC (N=238)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chilblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hodgkins's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Confusion state (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Toe amputation (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP0420 Plus SOC (N=247) | Placebo Plus SOC (N=238)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Anemia of chronic disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 11 (12) | 15 (15)
Generalized oedema (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Swelling face (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0)
Ischemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertransaminasemia (Hepatobiliary disorders) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 3 (3)
Sepsis shock (Infections and infestations) | 1 (1) | 2 (2)
Staphylococcal bacteremia (Infections and infestations) | 2 (2) | 0 (0)
Streptococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 3 (3)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter sepsis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypervolemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Ischemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 5 (5) | 7 (7)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8) | 7 (7)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 (31) | 26 (27)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (8)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (4)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organizing pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Hypotension (Vascular disorders) | 10 (11) | 8 (8)
Hypovolemic shock (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Trial H5 Protocol (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/63/NCT05780463/Prot_000.pdf
  • Study Protocol: Master Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05780463/Prot_001.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT05780463/SAP_002.pdf
  • Informed Consent Form (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT05780463/ICF_003.pdf